CLINICAL TRIAL: NCT06267534
Title: Effects of a Mindfulness-based Mobile Applications Program on Mental Health of Emergency Nurses Caring for COVID-19 Patients
Brief Title: Mindfulness-based Mobile Applications Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yu-Chien Huang (Other)
Responsible Party: Sponsor-Investigator, Yu-Chien Huang, Principal Investigator, Mackay Memorial Hospital
Organization: Mackay Memorial Hospital (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: YCH
Record Dates: First submitted 2023-10-20; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Cell Phone Use; Nurse; Mental Health
MeSH Terms: conditions — COVID-19; Cell Phone Use; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindfulness-based mobile applications program (Experimental): mindfulness-based mobile applications program. There are five audio files, listen to one audio file for two days.
  Interventions: Device: mindfulness-based mobile applications program
- NO intervention (No Intervention): The control group received no intervention, Scale exam was performed before and after the program in both groups at the same time.

INTERVENTIONS:
Device: mindfulness-based mobile applications program — Every two days is the same practice sound file, which must be practiced in order, so each sound file will be locked, for example: 9/9, 9/10 listen to the first sound file practice, 9/11, 9/12 listen to the second Practice with two sound files... and so on. After two days, the sound files will be automatically unlocked, and the subjects can continue to practice. The first ten days need to be practiced in order. From the eleventh day, each sound file will be unlocked. You can choose an audio file to practice, and the page will record the time and items of the practice, and you can also use text to record your experience after the practice
  Arms: mindfulness-based mobile applications program

SUMMARY:
The goal of this type of study: quasi-experimental clinical trial . The purpose of this study is to explore the effects of applying mindfulness-based mobile applications program to maintaining mental health of emergency nurses during providing care to COVID-19 patients. The main question[s] it aims to answer are:

1. To explore the effect of mindfulness-based mobile device-assisted program on care stress of emergency nurses caring for COVID-19 patients.
2. To explore the impact of mindfulness-based mobile device-assisted programs on the psychological distress of emergency nurses caring for COVID-19 patients.
3. To explore the impact of a mindfulness-based mobile device-assisted program on compassion fatigue in emergency nurses caring for COVID-19 patients.

Participants will Mindfulness-based mobile device is provided to experimental group as assistance for 2 weeks. In the contrary, no intervention measure was assigned in the control group. Scale exam was performed before and after the program in both groups at the same time.

DETAILED DESCRIPTION:
This study was a quasi-experimental study with two groups of pretest and posttest to facilitate sampling from the emergency room of Mackay Memorial Hospital. Emergency nurses at Taipei Mackay Memorial Hospital were in the experimental group, and emergency nurses at Tamsui Mackay Memorial Hospital were in the control group. These cases are expected to be accepted. There were 54 people in the experimental group and 54 people in the control group. The experimental group received a two-week mindfulness-based mobility device-assisted program. The program is a mobile application developed by researchers and designed for use on smartphones, tablets, and other mobile devices. The program content is facilitated and guided by certified instructors from the Center for Mindfulness (CFM) at the University of Massachusetts Medical School. Five suitable sound files were provided to guide subjects in practicing mindfulness. Each audio file is approximately 10 to 15 minutes in length. The control group did not take any intervention measures. The experimental group was tested on the scale before and after the program, and the control group was also measured at the same time. Research tools include the Nursing Stress Scale, Psychological Distress Scale, and Compassion Exhaustion Scale. The SPSS 20.0 software package was used for statistical analysis and processing of the data, and covariates were used to analyze the results. The findings will help improve mental health by reducing stress, psychological distress and compassion fatigue among emergency nurse practitioners caring for COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

Have a license to practice nurses; have worked in the medical center for more than three months; and are emergency clinical nurses who have experience in caring for COVID-19 nucleic acid test patients.

Exclusion Criteria:

The exclusion criteria were emergency clinical nurses who had received courses related to mindfulness training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 102 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
The impact of mindfulness-based mobile device assistance program on the care stress of emergency nursing staff caring for COVID-19 patients | Two weeks
  This study uses the "Nursing Stress Questionnaire under the COVID-19 Epidemic" as a measure of caregiving stress. The content includes five major aspects: worries about social isolation (10 questions), discomfort caused by protective equipment (8 questions), and infection control. Difficulties and anxiety (7 questions), burden of caring for patients (7 questions), and policy pressure (8 questions). The scoring method adopts a four-point Likert scale, ranging from no pressure (0 points) to severe pressure (3 points), a total of 40 questions, with a total score of 0-120 points. The higher the score, the greater the caregiving pressure.emergency nurses caring for COVID-19 patients
Effects of mindfulness-based mobile device assistance program on psychological distress among emergency nursing staff caring for COVID-19 patients | Two weeks
  This study used the "Short Form Health Scale" to measure the degree of psychological distress among caregivers caring for COVID-19 patients. There are five questions in the questionnaire, and the scoring method adopts a five-point Likert scale, ranging from not at all (0 points) to very good (4 points), with a total score of 0-20 points. The grading method is: a total score ≤ 5 is within the normal range, indicating good physical and mental adaptation; 6-9 is considered mild emotional distress; 10-14 is considered moderate emotional distress; and a score of 15 or above is severe emotional distress.
Effects of a mindfulness-based mobile device-assisted program on compassion fatigue among emergency nursing staff caring for COVID-19 patients | Two weeks
  The amount of compassion fatigue is measured using 23 questions of the Compassion Fatigue Self Test (CFST) developed by Figley (1995). Compassion fatigue is graded. Scores below 30 are classified as low risk; scores between 31 and 35 are classified as low risk. Medium risk; 36-40 is considered high risk; above 41 is considered extremely high risk

CONTACTS AND LOCATIONS:
Locations (1):
- Yu-Chien Huang, Taipei, Zhongzheng District, Taiwan

IPD SHARING:
Plan to Share IPD: No